CLINICAL TRIAL: NCT02768467
Title: A Prospective Randomized Controlled Trial of Buccal Mucosa Donor Site Healing With Tissue Matrix Placement
Brief Title: Buccal Mucosa Healing Trial With Tissue Matrix Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-00669
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Tissue Grafts
Keywords: Alloderm graft; Allograft; Buccal Mucosa

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tissue Matrix Graft Placement (Experimental): After the buccal mucosa is removed during reconstructive surgery, the wound is covered with an acellular tissue collagen matrix
  Interventions: Procedure: Tissue Matrix Graft Placement
- Without stitches (Active Comparator): After the buccal mucosa is removed during reconstructive surgery, no stitches will be used for the wound to heal.
  Interventions: Procedure: No Stitches

INTERVENTIONS:
Procedure: Tissue Matrix Graft Placement — Subject will receive a covering for the wound post buccal mucosa removal.
  Arms: Tissue Matrix Graft Placement
Procedure: No Stitches — Subject will not receive stitches post buccal mucosa removal.
  Arms: Without stitches

SUMMARY:
Prior studies have been performed to understand the optimal way to minimize the morbidity rate of buccal mucosa. While some studies have reported primary closure to be inferior to healing by secondary intention, this appears to be true for large defects greater than 2 cm in width. For small defects for which the wound can be closed without tension, the most recent study has shown improved pain outcomes in the immediate post-operative setting, although no difference is seen long term whether or not the wound was primarily closed. However, for larger defects, standard practice is to allow delayed healing by secondary intention.

The use of Alloderm graft placement for donor site coverage was first described in Armenakas' group. Alloderm is an acellular dermal lattice from human allograft skin. The only study to report the use of Alloderm failed to find a significant improvement in patient outcomes; however, very small defects were included in this study and the control group underwent primary closure, which has been shown to be inferior for large defects. Importantly, no increase in post-operative pain was noted, although there was some increased swelling reported. From experience, patients with moderate and large (>2 cm width) defects following buccal mucosa harvest benefit from Alloderm placement with decreased post-operative pain, more rapid resumption of normal diet and mouth function with no associated increase in morbidity of the procedure. This study aims to determine whether this is a reliable improvement in technique.

This study will clarify how the cheek heals after the buccal mucosa is removed during reconstructive surgery. Subjects will be randomized to either receive tissue collagen matrix or no stitches after the surgery. Subjects will be evaluated up to six months to determine if the outcomes of the tissue matrix graft are better for the subject.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Male
* Patients with clinically necessary buccal mucosal graft >2 cm
* Patients who are able to present for pre-operative and post-operative evaluations
* Patients who are able to comprehend and read English

Exclusion Criteria:

* History of oral cancer
* Severe cognitive impairments
* Unwilling or unable to follow procedures in protocol
* Contraindicated to participate for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Pain Level | Six months
  Measured by the Visual Analog Scale

SECONDARY OUTCOMES:
Time to Normal Eating | Six Months
  This is measured by time.
Presence of Swelling | Six Months
  This is measured by time
Mouth mobility | Six Months
  This is measured by time
Presence of Paresthesia | Six Months
  This is measured by time

CONTACTS AND LOCATIONS:
Overall Officials: Lee Zhao, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States